CLINICAL TRIAL: NCT01139658
Title: Observational Cohort Study on the Prevention of Venous Thromboembolic Events After Elective Orthopaedic Surgery in Patients Treated With PRADAXA
Brief Title: Prevention of Venous Thromboembolic Events After Elective Orthopaedic Surgery in Patients Treated With PRADAXA
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.102
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2013-11

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- All comers

SUMMARY:
Observational cohort study on the prevention of venous thromboembolic events after elective orthopaedic surgery for Total Knee Replacement or Total Hip Replacement iin patients treated with PRADAXA to evaluate the efficacy ant safety of Pradaxa in real-life conditions

ELIGIBILITY:
Inclusion criteria:

1. Patients treated with Pradaxa undergoing surgery for Total Knee Replacement or Total Hip Replacement
2. Patients 18 years of age or older at the time of recruitment

Exclusion criteria:

1. Patients presenting contraindication to prescription of Pradaxa
2. Patients in whom long term Anti vitamin K treatment is indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Demographic, medical and chirurgical characteristics
Sampling Method: Probability Sample
Enrollment: 1676 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (53):
- France (53):
  - Boehringer Ingelheim Investigational Site 30, Angers
  - Boehringer Ingelheim Investigational Site 41, Arles
  - Boehringer Ingelheim Investigational Site 40, Beauvais
  - Boehringer Ingelheim Investigational Site 2, Berck
  - Boehringer Ingelheim Investigational Site 25, Bordeaux
  - Boehringer Ingelheim Investigational Site 45, Boulogne-sur-Mer
  - Boehringer Ingelheim Investigational Site 13, Bruay-la-Buissière
  - Boehringer Ingelheim Investigational Site 42, Cahors
  - Boehringer Ingelheim Investigational Site 50, Castelnau-le-Lez
  - Boehringer Ingelheim Investigational Site 36, Chantilly
  - Boehringer Ingelheim Investigational Site 35, Châteaubernard
  - Boehringer Ingelheim Investigational Site 10, Châteaubriant
  - Boehringer Ingelheim Investigational Site 9, Clinique Des Maussins-Paris
  - Boehringer Ingelheim Investigational Site 44, Dole
  - Boehringer Ingelheim Investigational Site 3, Dracy-le-Fort
  - Boehringer Ingelheim Investigational Site 46, Haguenau
  - Boehringer Ingelheim Investigational Site 33, Illkirch-Graffenstaden
  - Boehringer Ingelheim Investigational Site 23, La Roche-sur-Yon
  - Boehringer Ingelheim Investigational Site 22, Lannion
  - Boehringer Ingelheim Investigational Site 27, Le Blanc Menil
  - Boehringer Ingelheim Investigational Site 31, Le Port-Marly
  - Boehringer Ingelheim Investigational Site 21, Libourne
  - Boehringer Ingelheim Investigational Site 5, Lille
  - Boehringer Ingelheim Investigational Site 19, Lyon
  - Boehringer Ingelheim Investigational Site 47, Marcq En Bareuil
  - Boehringer Ingelheim Investigational Site 12, Mâcon
  - Boehringer Ingelheim Investigational Site 28, Mérignac
  - Boehringer Ingelheim Investigational Site 26, Morlaix
  - Boehringer Ingelheim Investigational Site 48, Nancy
  - Boehringer Ingelheim Investigational Site 7, Nancy
  - Boehringer Ingelheim Investigational Site 8, Nice
  - Boehringer Ingelheim Investigational Site 11, Paris
  - Boehringer Ingelheim Investigational Site 17, Paris
  - Boehringer Ingelheim Investigational Site 6, Paris
  - Boehringer Ingelheim Investigational Site 24, Perpignan
  - Boehringer Ingelheim Investigational Site 49, Ploemeur
  - Boehringer Ingelheim Investigational Site 14, Poissy
  - Boehringer Ingelheim Investigational Site 39, Pontarlier
  - Boehringer Ingelheim Investigational Site 43, Pringy
  - Boehringer Ingelheim Investigational Site 15, Reims
  - Boehringer Ingelheim Investigational Site 20, Rennes
  - Boehringer Ingelheim Investigational Site 53, Saint Colombe Les Viennes
  - Boehringer Ingelheim Investigational Site 52, Saint-Georges-de-Didonne
  - Boehringer Ingelheim Investigational Site 4, Saint-Grégoire
  - Boehringer Ingelheim Investigational Site 18, Saint-Priest-en-Jarez
  - Boehringer Ingelheim Investigational Site 32, Saint-Priest-en-Jarez
  - Boehringer Ingelheim Investigational Site 51, Saint-Saulve
  - Boehringer Ingelheim Investigational Site 37, Saumur
  - Boehringer Ingelheim Investigational Site 34, Semur-en-Auxois
  - Boehringer Ingelheim Investigational Site 1, Strasbourg
  - Boehringer Ingelheim Investigational Site 38, Toulouse
  - Boehringer Ingelheim Investigational Site 29, Tourcoing
  - Boehringer Ingelheim Investigational Site 16, Villeneuve-sur-Lot

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Knee Replacement: Patients undergoing elective total knee replacement (TKR) received a dose of dabigatran etexilate; the administered treatment was based on usual practice in a real-life setting.
- Total Hip Replacement: Patients undergoing elective total hip replacement (THR) received a dose of dabigatran etexilate; the administered treatment was based on usual practice in a real-life setting.
Period: Overall Study
Arm/Group | Total Knee Replacement | Total Hip Replacement
Started | 747 | 929
Completed | 691 | 816
Not Completed | 56 | 113
Not completed — Adverse Event | 10 | 27
Not completed — Lack of Efficacy | 15 | 7
Not completed — Withdrawal by Subject | 2 | 4
Not completed — No documentation of treatment | 1 | 0
Not completed — Other | 28 | 75

BASELINE CHARACTERISTICS:
Population: Treated population included patients who took at least one dose of Pradaxa. One additional patient was excluded from the analysis as they were missing their date of first dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Knee Replacement | Total Hip Replacement | Total
Number analyzed (Participants) | 746 | 929 | 1675
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (9.5) | 67.8 (11.7) | 68.69 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 497 | 494 | 991
  Male | 249 | 435 | 684
Creatinine clearance [Mean (Standard Deviation); unit: mL/min] | 86.4 (29.6) | 85.1 (31.9) | 85.7 (30.9)
Weight [Mean (Standard Deviation); unit: kilogramm] | 79.6 (16.3) | 74.5 (15.6) | 76.8 (15.9)
Height [Mean (Standard Deviation); unit: cm] | 164.6 (9.1) | 166.8 (9.1) | 165.8 (9.1)
Participants with a Alanine Aminotransferase (ALT) of >2x normal upper limit [Number; unit: participants] | 29 | 40 | 69
Participants with at least one thromboembolic risk factor [Number; unit: participants] | 151 | 145 | 296
Participants with at least one cardiovascular risk factor [Number; unit: participants] | 543 | 586 | 1129
Participants with at least one concomitant disease [Number; unit: participants] | 176 | 203 | 379
Previous treatment [Number; unit: participants]
  NSAID | 402 | 509 | 911
  Aspirin | 83 | 79 | 162
  Clopidogrel | 12 | 15 | 27
  Amiodarone | 7 | 7 | 14
  Hydroquindin | 0 | 0 | 0
  Verapimil | 4 | 3 | 7
Current treatment [Number; unit: participants]
  NSAID | 92 | 125 | 217
  Aspirin | 56 | 45 | 101
  Clopidogrel | 5 | 3 | 8
  Amiodarone | 7 | 7 | 14
  Hydroquinidin | 0 | 0 | 0
  Verapamil | 4 | 3 | 7
Type of orthopedic surgery [Number; unit: participants] | 746 | 929 | 1675
Indication for the surgery [Number; unit: participants]
  Osteoarthritis | 701 | 818 | 1519
  Repair of existing prothesis | 24 | 42 | 66
  Osteonecrosis | 7 | 30 | 37
  Post-trauma | 6 | 19 | 25
  Inflammatory arthritis | 6 | 10 | 16
  Other | 2 | 9 | 11
Duration of the surgery [Mean (Standard Deviation); unit: minutes] | 80.8 (27.5) | 70.1 (28.6) | 74.9 (28.1)
Type of anesthesia [Number; unit: participants]
  General | 463 | 742 | 1205
  Spinal | 281 | 187 | 468
  Epidural | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Symptomatic Venous Thromboembolic Events
Description: Occurrence of symptomatic venous thromboembolic (VTE) events in patients treated with Pradaxa (dabigatran etexilate) after orthopaedic surgery (either Total Hip Replacement (THR) or Total Knee Replacement surgery (TKR)). Symptomatic VTE events were defined as a confirmed proximal or distal deep vein thrombosis (DVT) or a confirmed pulmonary embolism (PE).
Time Frame: 11 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
participants | 19 | 5

2. Primary Outcome: Occurrence of Major Bleeding Events
Description: Occurrence of major bleeding events (MBEs) in patients treated with Pradaxa (dabigatran etexilate) after orthopaedic surgery (either THR or TKR surgery). MBEs were defined as any fatal haemorrhage, any overt bleeding greater than could be expected combined with a loss of haemoglobin ≥ 2 g/dL or requiring transfusion ≥ 2 packed red blood cells units (PRBC), any symptomatic retroperitoneal, intracranial, intraocular or intraspinal haemorrhage or any bleeding requireing treatment cessation or reoperation.
  a confirmed proximal or distal deep vein thrombosis (DVT) or a confirmed pulmonary emboliam (PE).
Time Frame: 11 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
participants | 8 | 16

3. Secondary Outcome: Dosage of Pradaxa at Initiation
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
participants
  75 mg/day | 142 | 162
  110 mg/day | 394 | 417
  150 mg/day | 80 | 122
  220mg/day | 130 | 228

4. Secondary Outcome: Duration Between Surgery and First Dose of Pradaxa
Time Frame: 11 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
hours | 12.6 (14.5) | 14.6 (16.8)

5. Secondary Outcome: Duration of Treatment
Time Frame: 11 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
days | 27.5 (11.8) | 33.3 (10.4)

6. Secondary Outcome: Proportion of Patients With a Preoperative ALT Measurement
Time Frame: 11 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
percentage of participants | 73.3 | 74.5

7. Secondary Outcome: Adherence to Treatment
Description: The adherence to treatment was measured by patient declaration.
Time Frame: 11 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
percent | 98.6 (24.6) | 97.3 (24.6)

8. Secondary Outcome: Concomitant Treatments
Description: Concomitant treatments prescribed at hospital discharge.
Time Frame: 11 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
participants
  NSAID | 150 | 143
  Aspirin | 79 | 61
  Clopidogrel | 9 | 8
  Amiodarone | 7 | 6
  Hydroquinidin | 0 | 0
  Verapamil | 4 | 3

9. Secondary Outcome: Number of Patients Who Switched to Another Anticoagulant Therapy
Description: Treated population included patients who took at least one dose of Pradaxa. One additional patient was excluded from the analysis as they were missing their date of first dose.
Time Frame: 11 weeks
Measure: Number; unit: participants
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
participants | 43 | 45

10. Secondary Outcome: Prescription for the Surveillance of the Platelet Count on the Day of Hospital Discharge
Time Frame: 11 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
participants | 24 | 44

11. Secondary Outcome: Prescription for Nursing Care and Nurse Visits on the Day of Hospital Discharge
Time Frame: 11 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
participants | 420 | 584

12. Secondary Outcome: Reasons for Nurse Visits on the Day of Hospital Discharge
Time Frame: 11 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
participants
  Wound dressing care | 366 | 510
  Blood sample for platelet count | 27 | 69
  Other care | 29 | 54

13. Secondary Outcome: Frequency of Nurse Visits on the Day of Hospital Discharge
Time Frame: 11 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: times per week
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
times per week
  Wound dressing care | 2.3 (0.9) | 2.5 (0.9)
  Blood sample for platelet count | 1.7 (0.5) | 1.7 (0.5)

14. Secondary Outcome: Duration of Unplanned Hospitalizations at Visit 3
Time Frame: 11 weeks
Population: Outcome measure was not analyzed.
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Reasons for Unplanned Hospitalizations at Visit 3
Time Frame: 11 weeks
Population: Outcome measure was not analyzed.
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Reasons for Usual Follow-up
Time Frame: 11 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Total Knee Replacement | Total Hip Replacement
Number analyzed (Participants) | 746 | 929
participants
  Re-hospitalization | 11 | 17
  Consultation in the context of usual follow-up | 201 | 292
  Consultation outside the context of usual follow-u | 19 | 28

ADVERSE EVENTS:
Time Frame: 11 weeks
Arm/Group | Total Knee Replacement | Total Hip Replacement
Serious Adverse Events (participants affected / at risk) | 48/746 | 37/929
Other Adverse Events (participants affected / at risk) | 0/746 | 0/929
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Knee Replacement (N=746) | Total Hip Replacement (N=929)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 3
Cardiac failure (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1
Colonic stenosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Device dislocation (General disorders) | 1 | 2
Impaired healing (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 3
Femur fracture (Injury, poisoning and procedural complications) | 0 | 4
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 0 | 4
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 2 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Micturition disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 2
Patellectomy (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 17 | 6
Femoral artery occlusion (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 2
Haemodynamic instability (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 3 | 0
Phlebitis deep (Vascular disorders) | 1 | 1
Pulmonary embolism (Vascular disorders) | 4 | 2
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Data for the following secondary endpoints were not collected:

Medical appointments with a general practitioner or specialist at visit 3, Frequency of medical appointments at visit 3, Prescription received at visit 3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.